CLINICAL TRIAL: NCT03639571
Title: A Two-period, Multiple and Single Dose, Randomised, Double-blind, Placebo-controlled, Healthy Volunteer, Phase I Study to Assess Irritation, Sensitization and Adhesion of a Novel Ibuprofen 200 mg TEPI Medicated Plaster
Brief Title: Phase I Study to Assess Irritation, Sensitization and Adhesion of a Novel Ibuprofen 200 mg TEPI Medicated Plaster
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medherant Ltd (Industry)
Collaborators: Cooperative Clinical Drug Research and Development AG (CCDRD AG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MED-IBU-102
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (Experimental): Ibuprofen 200mg TEPI medicated plaster
  Interventions: Drug: Ibuprofen 200 mg TEPI Medicated Plaster
- Placebo (Placebo Comparator): Placebo TEPI Plaster
  Interventions: Other: Placebo TEPI Plaster

INTERVENTIONS:
Drug: Ibuprofen 200 mg TEPI Medicated Plaster — Ibuprofen 200 mg TEPI Medicated Plaster, manufactured by AdhexPharma, France on behalf of Medherant Ltd., UK
  Arms: Test
Other: Placebo TEPI Plaster — Placebo TEPI Plaster, manufactured by AdhexPharma, France on behalf of Medherant Ltd., UK
  Arms: Placebo

SUMMARY:
This trial will be conducted with the aim to investigate the dermal response (skin irritation, sensitization) and the adhesion of Ibuprofen 200 mg TEPI Medicated Plaster as compared to a Placebo TEPI Plaster in two phases:

Induction Phase: multiple dose application of one active and one placebo plaster on 5 consecutive days in which the plasters remain in place for 23 hours ± 30 min a day and Challenge Phase: single dose application of one active and one placebo plaster which remain in place for 48 hours ± 30 min.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subject
* Age between 18 and 65 years
* Physically and mentally healthy as judged by means of medical and standard laboratory examinations
* Non-smokers or ex-smokers (stopped at least 6 months ago) with a smoking history of ≤5 pack-year equivalents (1 pack-year equivalent is equal to smoking 1 pack per day for 1 year*****) and non-users of other nicotine containing products, confirmed by urine cotinine test
* Weight ≥ 60 kg and BMI within the range (including the borders) of 18.0 to 30.0 kg/m2
* Informed consent given in written form.

Exclusion Criteria:

* Participation in another clinical trial at same time or within the preceding 90 days (calculated from the date of the final examination of the previous study)
* Fertile women without reliable contraception method. List of allowed medically accepted contraceptive methods and the allowed HRT (used at least 4 weeks prior entry visit and not to be changed for the duration of the study):
* combination of 2 barrier methods: female/male condoms, diaphragms, spermicides
* intrauterine devices (IUD): inert or copper-releasing or progestinreleasing IUD
* hormonal methods: combined oestrogen/progestin injectable contraceptives, progestin only injectable contraceptives, Norplant implants, skin patches, NuvaRing®
* Hormone Replacement Therapy (HRT)
* voluntary sterilization (female tubal occlusion).
* Randomisation into the present trial more than once
* History of drug abuse or use of illegal drugs: use of soft drugs, e.g. marihuana within 6 months of screening or hard drugs, e.g. cocaine, amphetamines, phencyclidine within 1 year of screening
* Alcohol abuse, i.e. regular use of more than 2 units of alcohol per day or 10 units per week or a history of alcoholism (one unit of alcohol equals 250 ml beer, 125 ml wine or 25 ml spirits) or recovered alcoholics
* Positive drug screening and/or positive alcohol test at entry (screening) visit, or on Day -1, or on Day 19
* Pregnant and/or nursing women. Positive pregnancy test at entry (screening) visit, or on Day -1, or on Day 19
* Allergic diathesis or any clinically significant allergic disease (i.e. asthma or bronchial hyper-reactivity, contact dermatitis)
* Known allergy to sticking plaster or to the ingredients of the products
* Dermatologic disease that might interfere with the evaluation of test site reaction
* Active skin disease
* Subjects with tattoos, sunburn, coloration, open sores or scars on site of application
* Subject with excessive hair at site of plaster application
* Intake of systemic drugs interfering with the immune system (e.g. antiinflammatories, corticosteroids, immune-suppressants or antihistamines) within 2 weeks before and during the study
* Topical therapy with analgesics or corticosteroids or antihistamines at the application sites within 2 weeks before and during the study
* Intake or administration of any systemic or topical medication (including prescribed medication, OTC medication, and especially use of ointments, gels or patches for skin application) within 2 weeks before entry (screening) visit and during the study
* Use of topical products without medication at the application sites (including make-up, sunscreen, creams, lotions, powders, alcohol) from 7 days prior entry (screening) visit and during the study
* Intensive UV-light exposure (sunbath) at the application sites within 2 weeks before entry (screening) visit and during the study
* Use of tanning beds at the application sites within 2 weeks before entry (screening) visit and during the study
* Any method of hair removal (e.g. waxing, shaving, epilating, laser) at the application sites from 7 days before entry (screening) visit and during the study
* Presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, haematological, gastrointestinal, neurological, psychiatric or other diseases (e.g. autoimmune disorders such as lupus erythematosus)
* Clinically significant illness within 4 weeks before entry (screening) visit and during the study
* Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies [
* Systolic blood pressure outside the range of 100 to 140 mmHg and/or diastolic blood pressure outside the range of 60 to 90 mmHg12 at entry (screening) visit
* Heart rate outside the range of 50 to 90 beats/min at entry (screening) visit
* Respiratory rate outside the range of 12-24 breaths/min at entry (screening) visit
* Axillary body temperature outside the interval of 35.5 to 37.1°C at entry (screening) visit
* Any clinically significant abnormality of the resting ECG (12-lead) (i.e. AV block, 2° to 3°, sinus bradycardia, sick sinus syndrome, SA block)
* Laboratory values outside normal range with clinical relevance at entry (screening) examination
* Not fulfilling study specific restrictions and diet
* Subjects who are known or suspected:
* not to comply with the study directives
* not to be reliable or trustworthy
* not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed
* to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the inconvenience they may be involved in
* subject is a dependent person, e.g. a relative, family member, or member of the investigator's or sponsor's staff
* subject is in custody or submitted to an institution due to a judicial order.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Mean Irritation Score | 10 days
  Average of Dermal Response Scores Score Definition 0 - No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal oedema or minimal papular response
  3. - Erythema and papules
  4. - Definite oedema
  5. - Erythema, oedema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site
Total Cumulative Irritation Score | 10 dyas
  Sum of Dermal Response Scores - Score Definition 0 - No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal oedema or minimal papular response
  3. - Erythema and papules
  4. - Definite oedema
  5. - Erythema, oedema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site

SECONDARY OUTCOMES:
Mean Combined Dermal Response Score | 10 days
  Average of Dermal Response + Other Effects Score Dermal score - as explained above other effect score - Score Definition 0 - None observed
  1. - Slight glazed appearance
  2. - Marked glazing
  3. - Glazing with peeling and cracking
  4. - Glazing with fissures Film of dried serous exudates covering all or part of the plaster site Small petechial erosions and/or scabs
Total Combined Dermal Response Score | 10 days
  Sum of Dermal Response Score and Other Effects Score Dermal Response score - As explained above Other effects score - As explained above
Combined Dermal Response Scores | 10 days
  Combined Dermal Response Scores ≥2 Dermal response score - As explained above other effects score - as explained above

CONTACTS AND LOCATIONS:
Locations (1):
- MHAT, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No